CLINICAL TRIAL: NCT07186426
Title: A Multi-Center, Randomized, Double-Blind, Placebo/Active-Controlled Phase III Clinical Study to Evaluate the Efficacy and Safety of HSK21542 Injection for Postoperative Pain Treatment in Orthopedic Surgery
Brief Title: A Clinical Trial Evaluating the Efficacy and Safety of HSK21542 in Patients for Postoperative Pain Treatment in Orthopedic Surgery
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSK21542-305
Record Dates: First submitted 2025-09-04; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Postoperative Pain Management
MeSH Terms: interventions — Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HSK21542 (Experimental): Patients administrated with HSK21542
  Interventions: Drug: HSK21542
- Placebo control (Placebo Comparator): Patients administrated with placebo
  Interventions: Drug: Placebo
- Actice control (Active Comparator): Patients administrated with morphine
  Interventions: Drug: morphine

INTERVENTIONS:
Drug: HSK21542 — Patients administrated with HSK21542
  Arms: HSK21542
Drug: Placebo — Patients administrated with placebo
  Arms: Placebo control
Drug: morphine — Patients administrated with morphine
  Arms: Actice control

SUMMARY:
This is a multi-center, randomized, double-blind, placebo/active-controlled study. 405 subjects undergoing orthopedic surgery under general anesthesia are planned to be enrolled and randomized into the HSK21542 group, morphine group, and placebo group.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old ≤ age ≤70 years old, regardless of gender;
* 18 kg/m2≤BMI≤30 kg/m2，meet the weight range specified in the protocol；
* American Society of Anesthesiologists (ASA) grade ⅰ-ⅲ;
* Accept hip replacement under general anesthesia;
* Within 4 hours after the end of surgery, NRS≥4 in the resting state at any time;
* Fully understand and voluntarily participate this trial, and sign the informed consent form;

Exclusion Criteria:

* Patients with allergy to opioids or any component of the trial drug；
* Patients with a history of severe cardiovascular and cerebrovascular diseases, ,and psychiatric disorders;
* Last use of opioid or non-opioid analgesics less than 5 half-lives or the duration of drug efficacy prior to randomization; use of drugs with unclear half-lives that may affect analgesic efficacy within 7 days prior to randomization, or last use of drugs affecting analgesic efficacy less than 5 half-lives prior to randomization, as well as Chinese herbal medicines or proprietary Chinese medicines deemed by the investigator as potentially impacting the evaluation of efficacy and safety；
* Continuous use of opioid analgesics for more than 7 days for any reason within 30 days prior to screening;
* Laboratory test results during the screening period meeting any of the following criteria: 1) Significantly abnormal hematology results; 2) Significantly abnormal prothrombin time test results; 3) Significantly abnormal liver or kidney function; 4) Significantly abnormal fasting blood glucose;
* Positive test results during the screening period for hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCVAb), syphilis antibody, or human immunodeficiency virus (HIV) antibody;
* A history of drug, drug, and/or alcohol abuse；
* Participate in any clinical trail within 30 days;
* Pregnant or lactating female subjects；
* Subjects of childbearing potential who are unwilling to use contraception throughout the study period or plan to become pregnant within 3 months after the study.；
* Subjects with any other factor considered by the investigator to be ineligible for participation in the trial.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 405 (Estimated)
Dates: Start 2025-07-28 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Sum of Pain Intensity Differences (SPID) | 48 hours
  Sum of Pain Intensity Differences (SPID) of each group

SECONDARY OUTCOMES:
Proportion of subjects experiencing nausea | 48 hours
  Proportion of subjects experiencing nausea of each group
Proportion of subjects experiencing vomit | 48 hours
  Proportion of subjects experiencing vomit of each group
Sum of Pain Intensity Differences (SPID) in other time frame | 0-8 hours, 0-24 hours, 24-48 hours
  Sum of Pain Intensity Differences (SPID) in other time frame
Number of times rescue analgesic medications were administered. | 48 hours
  Number of times rescue analgesic medications were administered.
Total morphine consumption | 48 hours
  Total morphine consumption of each group

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Xuanwu Hospital Capital Medical University, Beijing, Beijing Municipality
  - Xiangya Hospital of Central South University, Changsha, Hunan

IPD SHARING:
Plan to Share IPD: No